CLINICAL TRIAL: NCT00775099
Title: The Effects of Combustion-Derived Air Pollution on Vascular Vasomotor and Fibrinolytic Function in Healthy Volunteers (Diesel Exposure)
Brief Title: Combustion Derived Air Pollution and Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: National Institute for Public Health and the Environment (RIVM) (Other Government)
Responsible Party: Professor David E Newby, University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 05/S1103/46
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Endothelial Dysfunction
Keywords: Air Pollution; Particles; Particulate Matter; Vascular function; Endothelial function; Thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Filtered Air Exposure (Experimental): 1 hour exposure to filtered air during intermittent exercise
  Interventions: Procedure: Forearm Vascular Study; Procedure: Badimon Chamber
- Diesel Exhaust Exposure (Experimental): 1 hour exposure to dilute diesel exhaust at a concentration of 300 µg/m3 during intermittent exercise
  Interventions: Procedure: Forearm Vascular Study; Procedure: Badimon Chamber
- Filtered Diesel Exposure (Experimental): 1 hour exposure to diesel exhaust with all particulates filtered out using teflon filter with intermittent exercise
  Interventions: Procedure: Forearm Vascular Study; Procedure: Badimon Chamber
- PALAS Exposure (Experimental): 1 hour exposure to pure carbon particles produced by PALAS generator during intermittent exercise
  Interventions: Procedure: Forearm Vascular Study; Procedure: Badimon Chamber

INTERVENTIONS:
Procedure: Forearm Vascular Study — Forearm venous occlusion plethysmography to measure forearm blood flow during intra-arterial infusion of the vasodilators Verapamil (10-100 µg/min), bradykinin (100-1000 pmol/min), sodium nitroprusside (2-8 µg/min) and Acetylcholine (5-20 mg/min).
  Other Names: BK; SNP; ACh
Procedure: Badimon Chamber — Ex-vivo assessment of thrombus formation using Badimon Chamber

SUMMARY:
Air pollution is a major cause of cardiovascular morbidity and mortality. The components of air pollution responsible and the mechanisms through which they might mediate these harmful effects remain only partially understood. The link between cardiovascular disease and air pollution is strongest for fine particulate matter. Fine particulate matter (PM) is produced from the combustion of fossil fuels with the most significant threat thought to be posed by small particles less than 10µm (PM 10) which can be inhaled into the lungs. We propose to identify the precise component of diesel exhaust that mediates the adverse cardiovascular effects using a carbon particle generator, and a particle concentrator. The aim of this study proposal is to assess the vascular effects of different types and components of air pollution in healthy subjects. We intend to test the hypotheses that:

1. Combustion derived nanoparticulate causes an acute impairment of endothelial vasomotor and fibrinolytic function in healthy volunteers.
2. Exposure to combustion derived air pollution is associated with increased thrombus formation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Current smokers
* Significant occupational exposure to air pollution
* History of lung disease
* Women of child-bearing potential
* Malignant arrhythmias
* Renal or hepatic failure
* Significant co-morbidity
* Systolic blood pressure >190 or <100 mmHg
* Previous history of blood dyscrasia
* Unable to tolerate the supine position
* Lack of informed consent
* Blood donation within last 3 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-09; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow measured by forearm venous occlusion plethysmography in response to infused vasodilators | 6-8 hours after exposure

SECONDARY OUTCOMES:
Ex-vivo thrombus formation assessed using the Badimon chamber | 6 hours after exposure
Arterial stiffness measured by radial artery tonometry | Before and after exposure
Heart rate and heart rate variability measured with 3 lead Holter electrographic monitors | During and for 24 hours after exposure
Blood pressure | During and after exposure and during forearm study
Plasma t-PA and PAI concentrations following infusion of bradykinin | During forearm study
Plasma inflammatory markers IL-6, TNF-alpha, IL-1 and hsCRP | Before and after exposure
Platelet monocyte binding as measured by flow cytometry | After the exposure

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas L Mills, MB BCh MRCP, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom

REFERENCES:
- [Background] Mills NL, Tornqvist H, Robinson SD, Gonzalez M, Darnley K, MacNee W, Boon NA, Donaldson K, Blomberg A, Sandstrom T, Newby DE. Diesel exhaust inhalation causes vascular dysfunction and impaired endogenous fibrinolysis. Circulation. 2005 Dec 20;112(25):3930-6. doi: 10.1161/CIRCULATIONAHA.105.588962. PMID 16365212
- [Derived] Langrish JP, Watts SJ, Hunter AJ, Shah AS, Bosson JA, Unosson J, Barath S, Lundback M, Cassee FR, Donaldson K, Sandstrom T, Blomberg A, Newby DE, Mills NL. Controlled exposures to air pollutants and risk of cardiac arrhythmia. Environ Health Perspect. 2014 Jul;122(7):747-53. doi: 10.1289/ehp.1307337. Epub 2014 Mar 25. PMID 24667535